CLINICAL TRIAL: NCT03851848
Title: Joints Mobilization Versus Myofascial Release on Diabetic Patients With Painful Heel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Afnan Alabdulaaly, Principal Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: plantar heel pain
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Foot; Plantar Fasciitis
Keywords: Myofascial release; Ankle and foot mobilization; Diabetic patients; plantar heel pain
MeSH Terms: conditions — Diabetic Foot; Fasciitis, Plantar | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint mobilization (JM) group (Experimental): The Maitland mobilization technique will target three main joints of the affected foot in order to facilitate major ankle and foot movements: (1) Talocrural joint Anterior-posterior (AP) mobilization will be performed to enhance ankle dorsiflexion ROM; (2) first metatarsal phalangeal joint (FMTP) AP glide will be performed to facilitate big toe extension ROM; (3) subtalar joint traction will be performed to increase both foot eversion and inversion ROM, and lateral glide will be performed to reinforce inversion ROM.
  Interventions: Other: Joint mobilization (JM)
- Myofascial release (MFR) group (Experimental): The MFR technique will be performed as a direct trigger point release followed by deep soft tissue release for the calf muscles (gastrocnemius and soleus) and the plantar fascia .
  Interventions: Other: Myofascial release (MFR)

INTERVENTIONS:
Other: Joint mobilization (JM) — Joint mobilization (JM) is a manual therapy to move the joint in a desired direction. It is commonly used for improving the joints' ROM and pain intensity, and to overcome joint restriction.
  Arms: Joint mobilization (JM) group
Other: Myofascial release (MFR) — Myofascial release (MFR) is a technique in which a slow, sustained pressure is applied to the restricted soft tissue in order to restore optimal length, reduce pain and improve function.
  Arms: Myofascial release (MFR) group

SUMMARY:
Diabetes mellitus (DM) increases stiffness and thickness of foot structures. This may alter the foot's biomechanics and increase plantar pressure distribution, mainly on the forefoot region. Presence of plantar heel pain (PHP) also may alter the foot's rollover mechanism and increase plantar loading in the forefoot as a protective mechanism of pain. The risk of diabetic ulcer formation increases with these restricted ankle range of motion (ROM) and increased foot plantar pressure that may present in DM patient with PHP.

The association that has been established previously between limited ankle ROM and PHP leads to a reasonable utilization of joint and soft tissue mobilization in treating diabetic patients with PHP. The aim of this study is to investigate the immediate and short-term effect of a single session of ankle and foot joint mobilization (JM) versus Myofascial release (MFR) on pain intensity, ankle ROM, foot plantar pressure, dynamic and static balance, and functional level of diabetic patients with PHP.

The findings of this study will help to understand the effect of these two interventions on diabetic patients with PHP in term of the previously mentioned parameters. This may guide the physiotherapists to choose the best available technique to treat DM patients with PHP, and that may help to reduce the risk of DM foot complications.

DETAILED DESCRIPTION:
It is a clinical experimental study of 46 controlled diabetic patients (type II) above 30 years with unilateral PHP who will present to physiotherapy screening clinic through the medical referral. The participants will be evaluated then distributed randomly to receive a single session of either JM or MFR followed by an immediate reassessment and a follow-up reassessment after 2 weeks. The assessment will include ankle ROM, pain intensity (visual analog scale), static balance (one leg stance test), dynamic balance (time up and go test), plantar pressure distribution, and functional level (lower extremity functional scale LEFS). Analysis of parametric data will be done using ANOVA for the repeated measure. LEFS score will be calculated using Mann-Whitney U test for nonparametric data. Alpha < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Controlled diabetic patients (type II)
2. aged above 30 years
3. presented with unilateral plantar heel pain that diagnosed based on the following criteria (pain located at the heel or plantar surface of the mid-foot, morning first steps pain, and increased pain on weight bearing after a period of rest ).

Exclusion Criteria:

1. ankle or foot deformity.
2. corticosteroids injection in the heel in the past 3 months.
3. neurological disorders, nerve entrapment in lower extremities or peripheral neuropathy (by 10-g monofilament and tuning fork of 128 Hz testing based on American Diabetes Association recommendations.
4. red flags to either the joints mobilization (JM) : (e.g. tumor, fracture, rheumatoid arthritis, osteoporosis, severe vascular disease, prolonged steroid use) or the myofascial release (MFR) (e.g. infective conditions) .

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity level will be measured using visual analog scale (VAS) | the change after 5 minutes of treatment and the change after 2 weeks of treatment .
  Pain level will be recorded using VAS. The VAS is a continuous and unidimensional scale that measures subjective pain intensity level. It is a line of 10 cm (100 mm) length, starting from zero, which indicates no pain, to ten that represents the maximum imaginable level of pain . The participants will be asked to record their current pain by drawing a perpendicular line to the VAS line at the point that reflects their pain level. The result will be scored by measuring the distance (mm) on 10-cm line between the zero and patient's mark using a ruler. For the scores interpretation, the higher scores indicate greater level of pain. VAS is a valid and reliable tool for measuring acute and chronic adult pain.
Talocrural joint dorsiflexion ROM will be measured using a universal goniometer | the change after 5 minutes of treatment and the change after 2 weeks of treatment .
  Talocrural joint dorsiflexion ROM will be measured using a universal goniometer. The patient will be in a supine position, with his foot hanging over the edge of the bed. The goniometer fulcrum will be placed on the lateral malleoli, the stationary arm in line with the fibular head, and the movable arm on the lateral border of the foot toward the fifth metatarsal head. The participant will be asked to move the ankle actively from the neutral position as far as possible toward dorsiflexion. It is a valid tool in measuring joints ROM and has a good intra-rater reliability in measuring ankle dorsiflexion . The ROM score will be expressed in degree.

SECONDARY OUTCOMES:
Functional level will be measured using Lower extremity functional scale (LEFS) | after 2 weeks of treatment .
  The participants' functional level will be measured using the Arabic version of LEFS. The scale is a self-report outcome measure that was established to assess the limitation of functional activity due to lower extremity musculoskeletal disorders. It consists of 20 questions, and each question is scored from zero (maximum difficulty or inability to perform the activity) to four (no difficulty). The maximum score is eighty, which represents the highest functional level. The minimal clinically important difference (MCID) is nine points. It is a valid tool and has excellent test-retest reliability in measuring activity limitation in patients with lower-extremity musculoskeletal disorders (that includes patient with plantar heel pain).
Static balance will be measured using One leg stance test (OLS) | the change after 5 minutes of treatment and the change after 2 weeks of treatment .
  The OLS test will be administered on the limb of PHP. The participant will stand on the affected side barefoot, both hands on the iliac crest and with both eyes closed. The patient's other leg will be slightly flexed off the ground. Verbal cue will be given to start the test; the participant will be asked to stand on the tested leg for as long as possible. The test will be finished either after completed 30 sec, or in these cases: when the standing foot moved or shifted, or when non-standing foot touch the ground . For the patient's safety, the therapist will be standing close to the patient throughout the test. .The test has a good Inter-rater reliability (ICC=0.75) and Inter-subject reliability (ICC=0.73)
Dynamic balance will be measured using Time up and go test (TUG) | the change after 5 minutes of treatment and the change after 2 weeks of treatment .
  The TUG test measures the ability of the participant to stand up from a standard armchair, walk for three meters, turn at a marked object and return back to the chair as fast as possible. The participant will receive a verbal command "go" to start the test. The timing will begin once the command is given and will stop once the patient return to the chair. To ensure the safety and prevent falls, the chair-back will be stabilized against the wall, the walking area will be free from obstacles, and the therapist will be close to the patient.The test has an excellent inter-rater (ICC=0.99) and test-retest (ICC=. 99) reliability
Foot plantar pressure distribution (FPP) will be measured using Platform Pedography system | the change after 5 minutes of treatment and the change after 2 weeks of treatment .
  Foot plantar pressure (FPP) will be evaluated using Platform Pedography system (EMED® system) . It consists of a platform that contains calibrated capacitive sensors and connected to the computer software operating system. The platform is inserted in the middle of a foamed walkway. The participant will be asked to stand barefoot on the platform with both arms held relaxed beside their trunk to assess the static foot pressure distribution. Then the patient will walk barefoot on the assessment-walking track with their regular speed and step length to evaluate the dynamic foot pressure distribution. The system is an accurate, valid and reliable tool for measuring static and dynamic foot pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Security Forces hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Celik D, Kus G, Sirma SO. Joint Mobilization and Stretching Exercise vs Steroid Injection in the Treatment of Plantar Fasciitis: A Randomized Controlled Study. Foot Ankle Int. 2016 Feb;37(2):150-6. doi: 10.1177/1071100715607619. Epub 2015 Sep 23. PMID 26400901
- [Background] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Background] Grieve R, Cranston A, Henderson A, John R, Malone G, Mayall C. The immediate effect of triceps surae myofascial trigger point therapy on restricted active ankle joint dorsiflexion in recreational runners: a crossover randomised controlled trial. J Bodyw Mov Ther. 2013 Oct;17(4):453-61. doi: 10.1016/j.jbmt.2013.02.001. Epub 2013 Apr 21. PMID 24139003
- [Background] Renan-Ordine R, Alburquerque-Sendin F, de Souza DP, Cleland JA, Fernandez-de-Las-Penas C. Effectiveness of myofascial trigger point manual therapy combined with a self-stretching protocol for the management of plantar heel pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2011 Feb;41(2):43-50. doi: 10.2519/jospt.2011.3504. Epub 2011 Jan 31. PMID 21285525